CLINICAL TRIAL: NCT02854280
Title: Brain During Effort : Effects of Hypoxia With Respiratory Patients
Acronym: NEUROX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC12.212
Record Dates: First submitted 2016-07-26; First posted 2016-08-03 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Sleep Apnea Obstructive (OSA); Healthy Volunteers
Keywords: Hypoxia; Brain; Effort
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chronic Obstructive Pulmonary Disease (COPD) (Active Comparator): 18 patients
  Interventions: Biological: Pedalling exercise on a cycle ergometer; Biological: Isolated contractions of the quadriceps
- Sleep Apnea Obstructive (OSA) (Active Comparator): 18 patients
  Interventions: Biological: Pedalling exercise on a cycle ergometer; Biological: Isolated contractions of the quadriceps
- Healthy Volunteers (Active Comparator): 36 control patients
  Interventions: Biological: Pedalling exercise on a cycle ergometer; Biological: Isolated contractions of the quadriceps

INTERVENTIONS:
Biological: Pedalling exercise on a cycle ergometer — At 80% of the maximal aerobic power, until exhaustion
Biological: Isolated contractions of the quadriceps — Until exhaustion

SUMMARY:
Brain oxygenation is determined by the product of CaO2 and the cerebral blood flow (CBF), the modification of one or the other can affect the neuronal O2 availability.

Besides the effect of the PaO2, the CBF is also regulated by the PaCO2. During effort in state of hypoxia, the drop of the PaO2 associated to a potential decrease of the PaCO2 and therefore of the CBF, can create an important dizziness between the demand and the supply of cerebral O2.

It seems that hypoxia can trouble in a significant way the response of central neurons, just as the production of a motor cortex generated motor command.

Studies suggest that exercise in severe hypoxia condition can constitute a necessary threat for brain oxygenation and the motor command, with the consequence a decrease of the exercise performance.

This projects aim to study effects of hypoxia on the brain function for patients suffering from chronic respiratory disease. Neurophysiologic responses of the brain while resting or exercising, including drip and cerebral oxygenation, cortical excitation and motor command resulting for hypoxic subjects before and after a treatment to correct abnormalities of gaz in blood.

The study will use a multidisciplinary and supplementary methodological approach : the near-infrared spectroscopy (NIRS) to appreciate the drip and cerebral oxygenation, CBF, neurostimulation procedures and electromyography (EMG) to appreciate the cortical excitability, measure the level of central activation and motor command.

The goals of this study will be :

* Measure the drip and cerebral oxygenation, the cortical excitability, mechanisms of voluntary activation and central fatigue to the effort for the chronic hypoxemic patient compared to healthy control subjects.
* Analyse disruptions of locomotion parameters and posturographyc, in simple and double task, involving different levels of cerebral task.
* Analyse acute effects of an improvement of arterial oxygenation for patients suffering from chronic obstructive pulmonary disease (COPD) on drip and cerebral oxygenation, cortical excitability, mechanisms of voluntary activation and central fatigue.
* Evaluate effects of a treatment by continuous positive airway pressure (CPAP) for patients suffering from obstructive sleep apnea (OSA) with the same parameters.

ELIGIBILITY:
Inclusion Criteria:

COPD patients

* stages GOLD III - IV, FEV1/FVC ratio < 0,7 and maximum voluntary ventilation (MVV) < 50% of predicted values
* BMI < 30 kg/m²
* Age between 18 and 80 years
* Non-smoking or ex-smoker (stop since more than 3 months)
* Stable condition since more than 3 months
* PaCO2 < 45 mmHg resting with ambiant air
* No OSA diagnostic

OSA patients

* Severe OSA recently dignosed (apnoea-Hypopnoea Index (AHI) > 30)
* Score on Epworth Sleepiness Scale (ESS) > 10
* Age between 18 and 80 years
* BMI < 30 kg/m²

Control subjects

* Age between 18 and 80 years
* BMI < 30 kg/m²
* Non-smoker
* Without any chronic respiratory pathology, cardiovascular, metabolic, renal or neuromuscular, vestibular and/or visual disorder

Exclusion Criteria:

OSA and COPD patients

* Pathologies cardiovascular, neuromuscular, métabolic, renal
* Alcoholism
* BMI > 30 kg/m²
* Psychiatric disorders or history of behavioural disorders, vision disorders, vestibular disorders, neurologic disease sensitive to disrupt the postural control and the walking, cognitive disorders
* Instability since less than 3 months
* Counter argument to the application of an external magnetic field

Control subjects

* Respiratory pathologies, cardiovascular, neuromuscular, metabolic, renal
* Alcoholism
* BMI > 30 kg/m²
* Psychiatric disorders or history of behavioural disorders
* Counter argument to the application of an external magnetic field

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Near-infrared spectroscopy (NIRS) | Half an hour
  Quantities of total desoxyhemoglobin and hemoglobin at muscular and cerebral levels while resting or during effort in response to inhalation of variable fractions of O2 and CO2.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Levy, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Ainslie PN, Poulin MJ. Ventilatory, cerebrovascular, and cardiovascular interactions in acute hypoxia: regulation by carbon dioxide. J Appl Physiol (1985). 2004 Jul;97(1):149-59. doi: 10.1152/japplphysiol.01385.2003. Epub 2004 Mar 5. PMID 15004003
- [Background] Amann M, Romer LM, Subudhi AW, Pegelow DF, Dempsey JA. Severity of arterial hypoxaemia affects the relative contributions of peripheral muscle fatigue to exercise performance in healthy humans. J Physiol. 2007 May 15;581(Pt 1):389-403. doi: 10.1113/jphysiol.2007.129700. Epub 2007 Feb 22. PMID 17317739
- [Background] ASTRAND PO, CUDDY TE, SALTIN B, STENBERG J. CARDIAC OUTPUT DURING SUBMAXIMAL AND MAXIMAL WORK. J Appl Physiol. 1964 Mar;19:268-74. doi: 10.1152/jappl.1964.19.2.268. No abstract available. PMID 14155294
- [Background] Barnes M, Goldsworthy UR, Cary BA, Hill CJ. A diet and exercise program to improve clinical outcomes in patients with obstructive sleep apnea--a feasibility study. J Clin Sleep Med. 2009 Oct 15;5(5):409-15. PMID 19961023
- [Background] Bassett DR Jr, Howley ET. Limiting factors for maximum oxygen uptake and determinants of endurance performance. Med Sci Sports Exerc. 2000 Jan;32(1):70-84. doi: 10.1097/00005768-200001000-00012. PMID 10647532
- [Background] Bedard MA, Montplaisir J, Richer F, Rouleau I, Malo J. Obstructive sleep apnea syndrome: pathogenesis of neuropsychological deficits. J Clin Exp Neuropsychol. 1991 Nov;13(6):950-64. doi: 10.1080/01688639108405110. PMID 1779033
- [Background] Beebe DW, Groesz L, Wells C, Nichols A, McGee K. The neuropsychological effects of obstructive sleep apnea: a meta-analysis of norm-referenced and case-controlled data. Sleep. 2003 May 1;26(3):298-307. doi: 10.1093/sleep/26.3.298. PMID 12749549
- [Background] Bergh U, Ekblom B, Astrand PO. Maximal oxygen uptake "classical" versus "contemporary" viewpoints. Med Sci Sports Exerc. 2000 Jan;32(1):85-8. doi: 10.1097/00005768-200001000-00013. PMID 10647533
- [Background] Bhambhani Y, Malik R, Mookerjee S. Cerebral oxygenation declines at exercise intensities above the respiratory compensation threshold. Respir Physiol Neurobiol. 2007 May 14;156(2):196-202. doi: 10.1016/j.resp.2006.08.009. Epub 2006 Aug 30. PMID 17045853
- [Background] Blomstrand E. Amino acids and central fatigue. Amino Acids. 2001;20(1):25-34. doi: 10.1007/s007260170063. PMID 11310928
- [Background] Brugniaux JV, Hodges AN, Hanly PJ, Poulin MJ. Cerebrovascular responses to altitude. Respir Physiol Neurobiol. 2007 Sep 30;158(2-3):212-23. doi: 10.1016/j.resp.2007.04.008. Epub 2007 May 1. PMID 17544954
- [Background] Calbet JA, Boushel R, Radegran G, Sondergaard H, Wagner PD, Saltin B. Why is VO2 max after altitude acclimatization still reduced despite normalization of arterial O2 content? Am J Physiol Regul Integr Comp Physiol. 2003 Feb;284(2):R304-16. doi: 10.1152/ajpregu.00156.2002. Epub 2002 Oct 3. PMID 12388462
- [Background] Canessa N, Castronovo V, Cappa SF, Aloia MS, Marelli S, Falini A, Alemanno F, Ferini-Strambi L. Obstructive sleep apnea: brain structural changes and neurocognitive function before and after treatment. Am J Respir Crit Care Med. 2011 May 15;183(10):1419-26. doi: 10.1164/rccm.201005-0693OC. Epub 2010 Oct 29. PMID 21037021
- [Background] Cannizzaro G, Garbin L, Clivati A, Pesce LI. Correction of hypoxia and hypercapnia in COPD patients: effects on cerebrovascular flow. Monaldi Arch Chest Dis. 1997 Feb;52(1):9-12. PMID 9151513
- [Background] Celli BR. Predictors of mortality in COPD. Respir Med. 2010 Jun;104(6):773-9. doi: 10.1016/j.rmed.2009.12.017. Epub 2010 Apr 22. PMID 20417082
- [Background] Chaudhuri A, Behan PO. Fatigue and basal ganglia. J Neurol Sci. 2000 Oct 1;179(S 1-2):34-42. doi: 10.1016/s0022-510x(00)00411-1. PMID 11054483
- [Background] Chien MY, Wu YT, Lee PL, Chang YJ, Yang PC. Inspiratory muscle dysfunction in patients with severe obstructive sleep apnoea. Eur Respir J. 2010 Feb;35(2):373-80. doi: 10.1183/09031936.00190208. Epub 2009 Jul 30. PMID 19643936
- [Background] Dalsgaard MK. Fuelling cerebral activity in exercising man. J Cereb Blood Flow Metab. 2006 Jun;26(6):731-50. doi: 10.1038/sj.jcbfm.9600256. PMID 16395281
- [Background] Davis JM, Alderson NL, Welsh RS. Serotonin and central nervous system fatigue: nutritional considerations. Am J Clin Nutr. 2000 Aug;72(2 Suppl):573S-8S. doi: 10.1093/ajcn/72.2.573S. PMID 10919962
- [Background] Foster GE, Hanly PJ, Ostrowski M, Poulin MJ. Effects of continuous positive airway pressure on cerebral vascular response to hypoxia in patients with obstructive sleep apnea. Am J Respir Crit Care Med. 2007 Apr 1;175(7):720-5. doi: 10.1164/rccm.200609-1271OC. Epub 2007 Jan 11. PMID 17218618
- [Background] Gonzalez-Alonso J, Dalsgaard MK, Osada T, Volianitis S, Dawson EA, Yoshiga CC, Secher NH. Brain and central haemodynamics and oxygenation during maximal exercise in humans. J Physiol. 2004 May 15;557(Pt 1):331-42. doi: 10.1113/jphysiol.2004.060574. Epub 2004 Mar 5. PMID 15004212
- [Background] Goodall S, Ross EZ, Romer LM. Effect of graded hypoxia on supraspinal contributions to fatigue with unilateral knee-extensor contractions. J Appl Physiol (1985). 2010 Dec;109(6):1842-51. doi: 10.1152/japplphysiol.00458.2010. Epub 2010 Sep 2. PMID 20813979
- [Background] Guezennec CY, Abdelmalki A, Serrurier B, Merino D, Bigard X, Berthelot M, Pierard C, Peres M. Effects of prolonged exercise on brain ammonia and amino acids. Int J Sports Med. 1998 Jul;19(5):323-7. doi: 10.1055/s-2007-971925. PMID 9721055
- [Background] Haddad GG, Jiang C. O2 deprivation in the central nervous system: on mechanisms of neuronal response, differential sensitivity and injury. Prog Neurobiol. 1993 Mar;40(3):277-318. doi: 10.1016/0301-0082(93)90014-j. No abstract available. PMID 7680137
- [Background] Hansen AJ. Effect of anoxia on ion distribution in the brain. Physiol Rev. 1985 Jan;65(1):101-48. doi: 10.1152/physrev.1985.65.1.101. No abstract available. PMID 3880896
- [Background] Herman T, Mirelman A, Giladi N, Schweiger A, Hausdorff JM. Executive control deficits as a prodrome to falls in healthy older adults: a prospective study linking thinking, walking, and falling. J Gerontol A Biol Sci Med Sci. 2010 Oct;65(10):1086-92. doi: 10.1093/gerona/glq077. Epub 2010 May 19. PMID 20484336
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Hopkinson NS, Sharshar T, Ross ET, Nickol AH, Dayer MJ, Porcher R, Jonville S, Moxham J, Polkey MI. Corticospinal control of respiratory muscles in chronic obstructive pulmonary disease. Respir Physiol Neurobiol. 2004 Jul 12;141(1):1-12. doi: 10.1016/j.resp.2004.04.003. PMID 15234671
- [Background] Ide K, Secher NH. Cerebral blood flow and metabolism during exercise. Prog Neurobiol. 2000 Jul;61(4):397-414. doi: 10.1016/s0301-0082(99)00057-x. PMID 10727781
- [Background] Jackson MJ. Molecular mechanisms of muscle damage. Mol Cell Biol Hum Dis Ser. 1993;3:257-82. doi: 10.1007/978-94-011-1528-5_10. No abstract available. PMID 8111542
- [Background] Jensen G, Nielsen HB, Ide K, Madsen PL, Svendsen LB, Svendsen UG, Secher NH. Cerebral oxygenation during exercise in patients with terminal lung disease. Chest. 2002 Aug;122(2):445-50. doi: 10.1378/chest.122.2.445. PMID 12171815
- [Background] Kayser B. Exercise starts and ends in the brain. Eur J Appl Physiol. 2003 Oct;90(3-4):411-9. doi: 10.1007/s00421-003-0902-7. Epub 2003 Jul 19. PMID 12883902
- [Background] Kayser B, Narici M, Binzoni T, Grassi B, Cerretelli P. Fatigue and exhaustion in chronic hypobaric hypoxia: influence of exercising muscle mass. J Appl Physiol (1985). 1994 Feb;76(2):634-40. doi: 10.1152/jappl.1994.76.2.634. PMID 8175572
- [Background] Kent-Braun JA. Central and peripheral contributions to muscle fatigue in humans during sustained maximal effort. Eur J Appl Physiol Occup Physiol. 1999 Jun;80(1):57-63. doi: 10.1007/s004210050558. PMID 10367724
- [Background] Lal C, Strange C, Bachman D. Neurocognitive impairment in obstructive sleep apnea. Chest. 2012 Jun;141(6):1601-1610. doi: 10.1378/chest.11-2214. PMID 22670023
- [Background] Lee M, Gandevia SC, Carroll TJ. Cortical voluntary activation can be reliably measured in human wrist extensors using transcranial magnetic stimulation. Clin Neurophysiol. 2008 May;119(5):1130-8. doi: 10.1016/j.clinph.2007.12.018. Epub 2008 Mar 4. PMID 18308630
- [Background] Lepers R, Maffiuletti NA, Rochette L, Brugniaux J, Millet GY. Neuromuscular fatigue during a long-duration cycling exercise. J Appl Physiol (1985). 2002 Apr;92(4):1487-93. doi: 10.1152/japplphysiol.00880.2001. PMID 11896014
- [Background] Levy P, Tamisier R, Minville C, Launois S, Pepin JL. Sleep apnoea syndrome in 2011: current concepts and future directions. Eur Respir Rev. 2011 Sep 1;20(121):134-46. doi: 10.1183/09059180.00003111. No abstract available. PMID 21881142
- [Background] Loeppky JA, Miranda FG, Eldridge MW. Abnormal cerebrovascular responses to CO2 in sleep apnea patients. Sleep. 1984;7(2):97-109. doi: 10.1093/sleep/7.2.97. PMID 6429811
- [Background] Macey PM, Henderson LA, Macey KE, Alger JR, Frysinger RC, Woo MA, Harper RK, Yan-Go FL, Harper RM. Brain morphology associated with obstructive sleep apnea. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1382-7. doi: 10.1164/rccm.200201-050OC. PMID 12421746
- [Background] Mayer P, Dematteis M, Pepin JL, Wuyam B, Veale D, Vila A, Levy P. Peripheral neuropathy in sleep apnea. A tissue marker of the severity of nocturnal desaturation. Am J Respir Crit Care Med. 1999 Jan;159(1):213-9. doi: 10.1164/ajrccm.159.1.9709051. PMID 9872841
- [Background] Mazza S, Pepin JL, Naegele B, Plante J, Deschaux C, Levy P. Most obstructive sleep apnoea patients exhibit vigilance and attention deficits on an extended battery of tests. Eur Respir J. 2005 Jan;25(1):75-80. doi: 10.1183/09031936.04.00011204. PMID 15640326
- [Background] Miscio G, Milano E, Aguilar J, Savia G, Foffani G, Mauro A, Mordillo-Mateos L, Romero-Ganuza J, Oliviero A. Functional involvement of central nervous system at high altitude. Exp Brain Res. 2009 Mar;194(1):157-62. doi: 10.1007/s00221-009-1729-1. Epub 2009 Feb 17. PMID 19221723
- [Background] Mohamed-Hussein AA, Hamed SA, Abdel-Hakim N. Cerebral cortical dysfunction in chronic obstructive pulmonary disease: role of transcranial magnetic stimulation. Int J Tuberc Lung Dis. 2007 May;11(5):515-21. PMID 17439674
- [Background] Morrell MJ, Twigg G. Neural consequences of sleep disordered breathing: the role of intermittent hypoxia. Adv Exp Med Biol. 2006;588:75-88. doi: 10.1007/978-0-387-34817-9_8. PMID 17089881
- [Background] Naegele B, Thouvard V, Pepin JL, Levy P, Bonnet C, Perret JE, Pellat J, Feuerstein C. Deficits of cognitive executive functions in patients with sleep apnea syndrome. Sleep. 1995 Jan;18(1):43-52. PMID 7761742
- [Background] Nielsen HB, Boushel R, Madsen P, Secher NH. Cerebral desaturation during exercise reversed by O2 supplementation. Am J Physiol. 1999 Sep;277(3):H1045-52. doi: 10.1152/ajpheart.1999.277.3.H1045. PMID 10484427
- [Background] Noakes TD. Physiological models to understand exercise fatigue and the adaptations that predict or enhance athletic performance. Scand J Med Sci Sports. 2000 Jun;10(3):123-45. doi: 10.1034/j.1600-0838.2000.010003123.x. PMID 10843507
- [Background] Noakes TD, Peltonen JE, Rusko HK. Evidence that a central governor regulates exercise performance during acute hypoxia and hyperoxia. J Exp Biol. 2001 Sep;204(Pt 18):3225-34. doi: 10.1242/jeb.204.18.3225. PMID 11581338
- [Background] Nybo L, Moller K, Pedersen BK, Nielsen B, Secher NH. Association between fatigue and failure to preserve cerebral energy turnover during prolonged exercise. Acta Physiol Scand. 2003 Sep;179(1):67-74. doi: 10.1046/j.1365-201X.2003.01175.x. PMID 12940940
- [Background] O'Donoghue FJ, Wellard RM, Rochford PD, Dawson A, Barnes M, Ruehland WR, Jackson ML, Howard ME, Pierce RJ, Jackson GD. Magnetic resonance spectroscopy and neurocognitive dysfunction in obstructive sleep apnea before and after CPAP treatment. Sleep. 2012 Jan 1;35(1):41-8. doi: 10.5665/sleep.1582. PMID 22215917
- [Background] Oliviero A, Corbo G, Tonali PA, Pilato F, Saturno E, Dileone M, Versace V, Valente S, Di Lazzaro V. Functional involvement of central nervous system in acute exacerbation of chronic obstructive pulmonary disease A preliminary transcranial magnetic stimulation study. J Neurol. 2002 Sep;249(9):1232-6. doi: 10.1007/s00415-002-0817-y. PMID 12242545
- [Background] Ozaki H, Watanabe S, Suzuki H. Topographic EEG changes due to hypobaric hypoxia at simulated high altitude. Electroencephalogr Clin Neurophysiol. 1995 May;94(5):349-56. doi: 10.1016/0013-4694(94)00311-8. PMID 7774521
- [Background] Papadelis C, Kourtidou-Papadeli C, Bamidis PD, Maglaveras N, Pappas K. The effect of hypobaric hypoxia on multichannel EEG signal complexity. Clin Neurophysiol. 2007 Jan;118(1):31-52. doi: 10.1016/j.clinph.2006.09.008. Epub 2006 Nov 7. PMID 17088101
- [Background] Perrey S. Non-invasive NIR spectroscopy of human brain function during exercise. Methods. 2008 Aug;45(4):289-99. doi: 10.1016/j.ymeth.2008.04.005. Epub 2008 Jun 6. PMID 18539160
- [Background] Rasmussen P, Dawson EA, Nybo L, van Lieshout JJ, Secher NH, Gjedde A. Capillary-oxygenation-level-dependent near-infrared spectrometry in frontal lobe of humans. J Cereb Blood Flow Metab. 2007 May;27(5):1082-93. doi: 10.1038/sj.jcbfm.9600416. Epub 2006 Nov 1. PMID 17077816
- [Background] Rasmussen P, Nielsen J, Overgaard M, Krogh-Madsen R, Gjedde A, Secher NH, Petersen NC. Reduced muscle activation during exercise related to brain oxygenation and metabolism in humans. J Physiol. 2010 Jun 1;588(Pt 11):1985-95. doi: 10.1113/jphysiol.2009.186767. Epub 2010 Apr 19. PMID 20403976
- [Background] Reichmuth KJ, Dopp JM, Barczi SR, Skatrud JB, Wojdyla P, Hayes D Jr, Morgan BJ. Impaired vascular regulation in patients with obstructive sleep apnea: effects of continuous positive airway pressure treatment. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1143-50. doi: 10.1164/rccm.200903-0393OC. Epub 2009 Sep 10. PMID 19745203
- [Background] Remsburg S, Launois SH, Weiss JW. Patients with obstructive sleep apnea have an abnormal peripheral vascular response to hypoxia. J Appl Physiol (1985). 1999 Sep;87(3):1148-53. doi: 10.1152/jappl.1999.87.3.1148. PMID 10484589
- [Background] Ries AL. Pulmonary rehabilitation: summary of an evidence-based guideline. Respir Care. 2008 Sep;53(9):1203-7. PMID 18718040
- [Background] Rupp T, Perrey S. Effect of severe hypoxia on prefrontal cortex and muscle oxygenation responses at rest and during exhaustive exercise. Adv Exp Med Biol. 2009;645:329-34. doi: 10.1007/978-0-387-85998-9_49. PMID 19227490
- [Background] Sassoon CS, Gruer SE, Sieck GC. Temporal relationships of ventilatory failure, pump failure, and diaphragm fatigue. J Appl Physiol (1985). 1996 Jul;81(1):238-45. doi: 10.1152/jappl.1996.81.1.238. PMID 8828670
- [Background] Sidhu SK, Bentley DJ, Carroll TJ. Locomotor exercise induces long-lasting impairments in the capacity of the human motor cortex to voluntarily activate knee extensor muscles. J Appl Physiol (1985). 2009 Feb;106(2):556-65. doi: 10.1152/japplphysiol.90911.2008. Epub 2008 Dec 4. PMID 19056999
- [Background] Subudhi AW, Dimmen AC, Roach RC. Effects of acute hypoxia on cerebral and muscle oxygenation during incremental exercise. J Appl Physiol (1985). 2007 Jul;103(1):177-83. doi: 10.1152/japplphysiol.01460.2006. Epub 2007 Apr 12. PMID 17431082
- [Background] Subudhi AW, Lorenz MC, Fulco CS, Roach RC. Cerebrovascular responses to incremental exercise during hypobaric hypoxia: effect of oxygenation on maximal performance. Am J Physiol Heart Circ Physiol. 2008 Jan;294(1):H164-71. doi: 10.1152/ajpheart.01104.2007. Epub 2007 Nov 21. PMID 18032522
- [Background] Szubski C, Burtscher M, Loscher WN. The effects of short-term hypoxia on motor cortex excitability and neuromuscular activation. J Appl Physiol (1985). 2006 Dec;101(6):1673-7. doi: 10.1152/japplphysiol.00617.2006. Epub 2006 Aug 10. PMID 16902059
- [Background] Szubski C, Burtscher M, Loscher WN. Neuromuscular fatigue during sustained contractions performed in short-term hypoxia. Med Sci Sports Exerc. 2007 Jun;39(6):948-54. doi: 10.1249/mss.0b013e3180479918. PMID 17545884
- [Background] Taylor JL, Allen GM, Butler JE, Gandevia SC. Supraspinal fatigue during intermittent maximal voluntary contractions of the human elbow flexors. J Appl Physiol (1985). 2000 Jul;89(1):305-13. doi: 10.1152/jappl.2000.89.1.305. PMID 10904066
- [Background] Teppema LJ, Dahan A. The ventilatory response to hypoxia in mammals: mechanisms, measurement, and analysis. Physiol Rev. 2010 Apr;90(2):675-754. doi: 10.1152/physrev.00012.2009. PMID 20393196
- [Background] Tuunanen PI, Kauppinen RA. Effects of oxygen saturation on BOLD and arterial spin labelling perfusion fMRI signals studied in a motor activation task. Neuroimage. 2006 Mar;30(1):102-9. doi: 10.1016/j.neuroimage.2005.09.021. Epub 2005 Oct 21. PMID 16243545
- [Background] Van de Ven MJ, Colier WN, Van der Sluijs MC, Kersten BT, Oeseburg B, Folgering H. Ventilatory and cerebrovascular responses in normocapnic and hypercapnic COPD patients. Eur Respir J. 2001 Jul;18(1):61-8. doi: 10.1183/09031936.01.00087501. PMID 11510807
- [Background] van de Ven MJ, Colier WN, van der Sluijs MC, Oeseburg B, Vis P, Folgering H. Effects of acetazolamide and furosemide on ventilation and cerebral blood volume in normocapnic and hypercapnic patients with COPD. Chest. 2002 Feb;121(2):383-92. doi: 10.1378/chest.121.2.383. PMID 11834647
- [Background] Verges S, Maffiuletti NA, Kerherve H, Decorte N, Wuyam B, Millet GY. Comparison of electrical and magnetic stimulations to assess quadriceps muscle function. J Appl Physiol (1985). 2009 Feb;106(2):701-10. doi: 10.1152/japplphysiol.01051.2007. Epub 2008 Aug 28. PMID 18756009
- [Background] Vivodtzev I, Flore P, Levy P, Wuyam B. Voluntary activation during knee extensions in severely deconditioned patients with chronic obstructive pulmonary disease: benefit of endurance training. Muscle Nerve. 2008 Jan;37(1):27-35. doi: 10.1002/mus.20867. PMID 17912747
- [Background] Volianitis S, Fabricius-Bjerre A, Overgaard A, Stromstad M, Bjarrum M, Carlson C, Petersen NT, Rasmussen P, Secher NH, Nielsen HB. The cerebral metabolic ratio is not affected by oxygen availability during maximal exercise in humans. J Physiol. 2008 Jan 1;586(1):107-12. doi: 10.1113/jphysiol.2007.142273. Epub 2007 Oct 11. PMID 17932151
- [Background] Wagner PD. Reduced maximal cardiac output at altitude--mechanisms and significance. Respir Physiol. 2000 Mar;120(1):1-11. doi: 10.1016/s0034-5687(99)00101-2. PMID 10786640
- [Background] Westerblad H, Allen DG, Bruton JD, Andrade FH, Lannergren J. Mechanisms underlying the reduction of isometric force in skeletal muscle fatigue. Acta Physiol Scand. 1998 Mar;162(3):253-60. doi: 10.1046/j.1365-201X.1998.0301f.x. PMID 9578370
- [Background] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181
- [Background] Yogev-Seligmann G, Hausdorff JM, Giladi N. The role of executive function and attention in gait. Mov Disord. 2008 Feb 15;23(3):329-42; quiz 472. doi: 10.1002/mds.21720. PMID 18058946
- [Derived] Marillier M, Gruet M, Baillieul S, Wuyam B, Tamisier R, Levy P, Pepin JL, Verges S. Impaired cerebral oxygenation and exercise tolerance in patients with severe obstructive sleep apnea syndrome. Sleep Med. 2018 Nov;51:37-46. doi: 10.1016/j.sleep.2018.06.013. Epub 2018 Jul 4. PMID 30099350